CLINICAL TRIAL: NCT06385197
Title: Improving the Effect of Dimethyl Fumarate and Diroximel Fumarate (DRF) for Patients With Multiple Sclerosis by Chronobiology
Brief Title: Improving the Effect of Multiple Sclerosis Drugs by Chronobiology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 170886-HMO-CTIL
Record Dates: First submitted 2024-04-17; First posted 2024-04-25 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: A controlled-randomization dosing regimen administered to patients with MS and provided by a designated app. The treatment limitations of time interval is pre-defined according to approved therapeutic windows.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients using the app for dosing regimen (Experimental): All of the enrolled patients will receive their dimethyl fumarate prescribed by their GP. During the 12 weeks' study period, patients in the intervention arm will receive the medication timed by the app- dose and time of administration will be determined using a designated app. The app will implement random changes in time of administration limited by a pre-defined range assigned by the therapeutic windows
  Interventions: Device: App randomizing dosing regimen

INTERVENTIONS:
Device: App randomizing dosing regimen — patients will receive their dimethyl fumarate treatment and the dose and time of administration will be determined using a designated app.

SUMMARY:
A trial for evaluating the ability to improve the effect of dimethyl fumarate in patients with Multiple Sclerosis (MS) by chronobiology A controlled-randomization dosing regimen administered to patients with MS and provided by a designated app. The treatment limitations of time interval is pre-defined according to approved therapeutic windows.

DETAILED DESCRIPTION:
Dimethyl fumarate (DMF) is an oral option for patients with relapsing forms of MS. The effectiveness of DMF on the clinical and radiological activity of multiple sclerosis were demonstrated in a real-world setting, both in naive patients and in those switching from other multiple sclerosis therapies. Sustained safety and efficacy of DMF was observed in patients continuing on treatment for up to 11 years, supporting DMF as a long-term treatment option for patients with MS. It continues to be an efficacious treatment for multiple sclerosis with a favorable safety profile demonstrated over 10 years of clinical use Patients who have partial response or non-responders in most cases require different medications associated with a less favorable safety profile. Recently fda approved Diroximel fumarate (DRF) is a noval drug which is bioequivalent to DMF regarding efficacy and safety profiles, differing only by chemical precursor structure which is hypothesized to elicit less irritation in the GI tract than DMF. Both drug active metabolites are similar in bioactivity and efficacy treating MS Many aspects of cellular physiology display circadian (approximately 12-h) rhythms. Dysfunction of the circadian clock molecular circuitry is associated with human health derangements, including neurodegeneration, increased risk of cancer, cardiovascular diseases and the metabolic syndrome. Recent evidences support a link between the circadian clock circuitry and biological cycles in multiple systems. Regular dosing of therapy may lead to compensatory mechanisms and are associated with adaptation of the immune system that may prohibit a maximal clinical effect.

This open-label study will test the implementation of controlled randomization of time of administration of Dimethyl fumarate to patients with MS. Random changes in the time of administration and dosages of Dimethyl fumarate within pre-defined approved limits which are within the approved therapeutic window will be provided to patient by a designated cellular application. Patients will be followed for 12 weeks for clinical improvement using the Expanded Disability Status Scale (EDSS) and MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-60 at the time of enrollment
2. A diagnosis of MS and treatment with dimethyl fumarateDimethyl fumarate or Diroximel fumarate for at least 6 months
3. Females of childbearing potential must be non-pregnant (as determined by a serum pregnancy test at enrollment) and agree to use adequate contraceptive means throughout the study.
4. Patients must be able to adhere to the visit schedule and protocol requirements and be available to complete the study.
5. Patients must satisfy a medical examiner about their fitness to participate in the study.
6. Patients must provide written informed consent to participate in the study.

Exclusion Criteria:

* 1. Active malignancy or any malignancy diagnosed in the last 5 years or previous diagnosis of hepatocellular carcinoma at any time.

  2. Known human deficiency virus (HIV) or Hepatitis virus infections. 3. The use of steroids, or other immunosuppression. 4. Participation in another clinical trial within 30 days prior to intervention.

  5. Patients with an inability to communicate well with the PI and staff (i.e., language problem, poor mental development or impaired cerebral function).

  6. Patients who will be unavailable for the duration of the trial, are likely to be noncompliant with the protocol, or who are felt to be unsuitable by the PI for any other reason.

  7. Any underlying medical condition that in the opinion of the study investigator impair the ability of the patient to complete the follow-up or to receive the planned treatment regimen

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-05-08 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
safety assessment | 12 weeks
  The primary outcome is to assess to assess the safety of incorporating controlled randomization to Dimethyl fumarate dosing regimen provided by an app in patients with MS. Safety will be assessed through clinical follow-up which will include history taking with emphasize on possible AE
assessment of AE | 12 weeks
  physical examination and assessment by EDSS score
assessment of AE | 12 weeks
  laboratory tests - detect changes in cbc for lymphopenia (below 1.03 10e9/L)

CONTACTS AND LOCATIONS:
Overall Officials: yoav hershkovtiz, md, Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gold R, Arnold DL, Bar-Or A, Fox RJ, Kappos L, Chen C, Parks B, Miller C. Safety and efficacy of delayed-release dimethyl fumarate in patients with relapsing-remitting multiple sclerosis: 9 years' follow-up of DEFINE, CONFIRM, and ENDORSE. Ther Adv Neurol Disord. 2020 May 12;13:1756286420915005. doi: 10.1177/1756286420915005. eCollection 2020. PMID 32426039
- [Background] Chinea A, Amezcua L, Vargas W, Okai A, Williams MJ, Su R, Parks B, Mendoza JP, Lewin JB, Jones CC. Real-World Safety and Effectiveness of Dimethyl Fumarate in Hispanic or Latino Patients with Multiple Sclerosis: 3-Year Results from ESTEEM. Neurol Ther. 2020 Dec;9(2):495-504. doi: 10.1007/s40120-020-00192-6. Epub 2020 May 29. PMID 32472385
- [Background] Barros A, Sequeira J, de Sousa A, Parra J, Brum M, Pedrosa R, Capela C. Real-Word Effectiveness and Safety of Dimethyl Fumarate in a Multiple Sclerosis Portuguese Population. Clin Neuropharmacol. 2020 May/Jun;43(3):55-60. doi: 10.1097/WNF.0000000000000391. PMID 32384308
- [Background] Lanzillo R, Moccia M, Palladino R, Signoriello E, Carotenuto A, Maniscalco GT, Sacca F, Bonavita S, Russo CV, Iodice R, Petruzzo M, Sinisi L, De Angelis M, Lavorgna L, De Rosa A, Romano F, Orlando V, Ronga B, Florio C, Lus G, Brescia Morra V. Clinical predictors of Dimethyl Fumarate response in multiple sclerosis: a real life multicentre study. Mult Scler Relat Disord. 2020 Feb;38:101871. doi: 10.1016/j.msard.2019.101871. Epub 2019 Nov 25. PMID 31786463
- [Background] Miclea A, Leussink VI, Hartung HP, Gold R, Hoepner R. Safety and efficacy of dimethyl fumarate in multiple sclerosis: a multi-center observational study. J Neurol. 2016 Aug;263(8):1626-32. doi: 10.1007/s00415-016-8175-3. Epub 2016 Jun 3. PMID 27260297
- [Background] Goldberger AL. Non-linear dynamics for clinicians: chaos theory, fractals, and complexity at the bedside. Lancet. 1996 May 11;347(9011):1312-4. doi: 10.1016/s0140-6736(96)90948-4. No abstract available. PMID 8622511
- [Background] Singh N, Moneghetti KJ, Christle JW, Hadley D, Plews D, Froelicher V. Heart Rate Variability: An Old Metric with New Meaning in the Era of using mHealth Technologies for Health and Exercise Training Guidance. Part One: Physiology and Methods. Arrhythm Electrophysiol Rev. 2018 Aug;7(3):193-198. doi: 10.15420/aer.2018.27.2. PMID 30416733
- [Background] Shields RW Jr. Heart rate variability with deep breathing as a clinical test of cardiovagal function. Cleve Clin J Med. 2009 Apr;76 Suppl 2:S37-40. doi: 10.3949/ccjm.76.s2.08. PMID 19376980
- [Background] Konig N, Singh NB, Baumann CR, Taylor WR. Can Gait Signatures Provide Quantitative Measures for Aiding Clinical Decision-Making? A Systematic Meta-Analysis of Gait Variability Behavior in Patients with Parkinson's Disease. Front Hum Neurosci. 2016 Jun 30;10:319. doi: 10.3389/fnhum.2016.00319. eCollection 2016. PMID 27445759
- [Background] Nayyar S, Hasan MA, Roberts-Thomson KC, Sullivan T, Baumert M. Effect of Loss of Heart Rate Variability on T-Wave Heterogeneity and QT Variability in Heart Failure Patients: Implications in Ventricular Arrhythmogenesis. Cardiovasc Eng Technol. 2017 Jun;8(2):219-228. doi: 10.1007/s13239-017-0299-9. Epub 2017 Mar 3. PMID 28258544
- [Background] Moon Y, Sung J, An R, Hernandez ME, Sosnoff JJ. Gait variability in people with neurological disorders: A systematic review and meta-analysis. Hum Mov Sci. 2016 Jun;47:197-208. doi: 10.1016/j.humov.2016.03.010. Epub 2016 Mar 26. PMID 27023045
- [Background] Moon Y, Sung J, An R, Hernandez ME, Sosnoff JJ. Gait variability in people with neurological disorders: A systematic review and meta-analysis. Hum Mov Sci. 2016;47:197-208. 14. Leino AD, King EC, Jiang W, et al. Assessment of tacrolimus intrapatient variability in stable adherent transplant recipients: Establishing baseline values. Am J Transplant. 2018. 15. Gueta I, Markovits N, Yarden-Bilavsky H, et al. High tacrolimus trough level variability is associated with rejections after heart transplant. Am J Transplant. 2018;18(10):2571-2578. 16. Gueta I, Markovits N, Yarden-Bilavsky H, et al. Intrapatient variability in tacrolimus trough levels after solid organ transplantation varies at different postoperative time periods. Am J Transplant. 2018. 17. Del Bello A, Congy-Jolivet N, Danjoux M, et al. High tacrolimus intra-patient variability is associated with graft rejection, and de novo donor-specific antibodies occurrence after liver transplantation. World J Gastroenterol. 2018;24(16):1795-1802. 18. Contin M, Alberghini L, Candela C, Benini G, Riva R. Intrapatient variation in antiepileptic drug plasma concentration after generic substitution vs stable brand-name drug regimens. Epilepsy Res. 2016;122:79-83. 19. Elgart V, Lin JR, Loscalzo J. Determinants of drug-target interactions at the single cell level. PLoS Comput Biol. 2018;14(12):e1006601. 20. Niederer SA, Lumens J, Trayanova NA. Computational models in cardiology. Nat Rev Cardiol. 2019;16(2):100-111. 21. Ilan Y. Overcoming Compensatory Mechanisms toward Chronic Drug Administration to Ensure Long-Term, Sustainable Beneficial Effects. Mol Ther Methods Clin Dev. 2020;18:335-344. 22. Kyriazis M. Practical applications of chaos theory to the modulation of human ageing: nature prefers chaos to regularity. Biogerontology. 2003;4(2):75-90. 23. Kessler A, Weksler-Zangen S, Ilan Y. Role of the Immune System and the Circadian Rhythm in the Pathogenesis of Chronic Pancreatitis: Establishing a Personalized Signature for Improving the Effect of Immunotherapies for Chronic Pancreatitis. Pancreas. 2020;49(8):1024-1032. 24. Potruch A, Khoury ST, Ilan Y. The role of chronobiology in drug-resistance epilepsy: The potential use of a variability and chronotherapy-based individualized platform for improving the response to anti-seizure drugs. Seizure. 2020;80:201-211. 25. Khoury T, Ilan Y. Introducing Patterns of Variability for Overcoming Compensatory Adaptation of the Immune System to Immunomodulatory Agents: A Novel Method for Improving Clinical Response to Anti-TNF Therapies. Front Immunol. 2019;10:2726. 26. Khoury T, Ilan Y. Introducing Patterns of Variability for Overcoming Compensatory Adaptation of the Immune System to Immunomodulatory Agents: A Novel Method for Improving Clinical Response to Anti-TNF Therapies. Frontiers in immunology. 2019;10:2726-2726. 27. Gelman R, Bayatra A, Kessler A, Schwartz A, Ilan Y. Targeting SARS-CoV-2 receptors as a means for reducing infectivity and improving antiviral and immune response: an algorithm-based method for overcoming resistance to antiviral agents. Emerg Microbes Infect. 2020;9(1):1397-1406.